CLINICAL TRIAL: NCT06818851
Title: The Effects of Henagliflozin on glucOse fLuctuation and Immunosenescence in Type 2 Diabetes pAtients on Insulin therapY: a Multicenter, Randomized, Double-blind, Placebo-controlled Study (the HOLIDYA Study)
Brief Title: The Effects of Henagliflozin on Glucose Fluctuation and Immunosenescence in Type 2 Diabetes Patients on Insulin Therapy
Acronym: HOLIDYA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: XH-24-011
Record Dates: First submitted 2025-01-23; First posted 2025-02-11 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Sodium-glucose cotransporter 2; glycemic variability; immunosenescence
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Henggliflozin 10mg per day for 16 weeks
  Interventions: Drug: Henggliflozin
- Control Group (Placebo Comparator): Placebo 10mg per day for 16 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Henggliflozin — Upon enrollment, at Visit 1 (baseline), overnight fasting blood and urine samples will be collected, and glucose levels will be monitored for 3-5 days using a continuous glucose monitoring (CGM) system (Medtronic MiniMed). After the preliminary assessment, participants will receiveHenggliflozin 10 mg once daily by oral administration for up to 16 weeks.
  Arms: Experimental Group
Other: Placebo — Upon enrollment, at Visit 1 (baseline), overnight fasting blood and urine samples will be collected, and glucose levels will be monitored for 3-5 days using a continuous glucose monitoring (CGM) system (Medtronic MiniMed). After the preliminary assessment, participants will receive a placebo once daily by oral administration for up to 16 weeks.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn if SGLT2 inhibitor Henggliflozin works to improve glucose variability in type 2 diabetes and if Henggliflozin can benefit immunosenescence.

The main questions it aims to answer are:

Does Henggliflozin as an add on treatment works to improve blood glucose fluctuation in type 2 diabetes? Does Henggliflozin has extra benefits like improve immunosenescence beyond hypoglycemic effects? Researchers will compare Henggliflozin to a placebo to see if Henggliflozin can improve glucose variability and immunosenescence.

Participants will:

Take Henggliflozin or a placebo every day for 16 weeks. Receive weekly follow-up calls to guide them in adjusting their insulin doses. Return for an on-site visit at 4 weeks and 16 weeks. Take a continuous glucose monitoring (CGM) for 7 days at the Visit 1 and at the end of the study.

DETAILED DESCRIPTION:
With the rising prevalence of diabetes, complications associated with the disease are becoming a significant threat to human health. The primary goal of diabetes treatment is to delay the onset of macrovascular and microvascular complications and to reduce cardiovascular disease (CVD)-related mortality. Numerous clinical studies have explored the relationship between glycemic variability (GV) and the risk of macrovascular disease. Recent research has shown that GV is closely associated with endothelial cell damage, which represents an early stage of atherosclerosis and serves as a predictive factor for CVD.

The mean amplitude of glycemic excursions (MAGE), a marker of daily GV related to postprandial hyperglycemia or hypoglycemia, is a critical determinant of the severity of coronary artery disease and an independent predictor of mortality risk. Over the long term, reducing daily GV can help lower cardiovascular events and mitigate cognitive decline in patients. Therefore, controlling GV is particularly important in reducing the risk of cardiovascular disease.

While there is no strong evidence yet to suggest that suppressing GV can directly reverse cardiovascular events, some studies indicate that antidiabetic medications that reduce GV can improve surrogate markers of cardiovascular risk factors. Sodium-glucose cotransporter 2 (SGLT2) inhibitors lower blood glucose by promoting glucose excretion through urine. Research has demonstrated that SGLT2 inhibitors can reduce cardiovascular risks; however, studies on their effect in suppressing GV remain insufficient.

This study is a multicenter, randomized, double-blind controlled trial aiming to enroll 64 participants with type 2 diabetes.

Eligible participants will be randomly assigned to one of two groups in a 1:1 ratio:

* Henggliflozin Group (n=32): Henggliflozin 10 mg, once daily.
* Placebo Control Group (n=32): Placebo, once daily.

Upon enrollment, at Visit 1 (baseline), overnight fasting blood and urine samples will be collected, and glucose levels will be monitored for 3-5 days using a continuous glucose monitoring (CGM) system. After the preliminary assessment, participants will receive either Henggliflozin 10 mg or a placebo once daily by oral administration for up to 16 weeks.

During the treatment period, weekly follow-up calls will be conducted to guide participants in adjusting their insulin doses until fasting blood glucose (FBG) reaches the target level (<7 mmol/L). Participants will return for an on-site visit at 4 weeks, during which medications will be retrieved, and relevant information recorded. Other antidiabetic medications, such as metformin, sulfonylureas, glinides, thiazolidinediones, or α-glucosidase inhibitors, may continue to be used at unchanged doses throughout the study. Participants will be encouraged to maintain their dietary and exercise regimens. If there is a risk of hypoglycemia, insulin doses may be reduced.

At the end of the 16-week treatment period, medications will be retrieved again, and fasting blood and urine samples will be collected. Glucose monitoring will be repeated using the CGM system. A safety follow-up call will be conducted two weeks after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus (T2DM) for at least 6 months based on the 1999 WHO criteria.

  * Age between 50 and 70 years at the time of signing the informed consent form (inclusive).
  * Poor glycemic control despite treatment with basal insulin or insulin degludec/aspart (with or without oral antidiabetic drugs) within the 3 months prior to screening.
  * HbA1c level above 8%.
  * BMI ≥ 20 kg/m².
  * C-peptide levels within the normal reference range.
  * Able to maintain stable dietary and exercise habits during the study.
  * Capable of understanding the study procedures and methods, willing to strictly comply with the clinical trial protocol, and voluntarily sign the informed consent form.

Exclusion Criteria:

* Patients considered by the investigator to have potential allergies to the components of the study drug or drugs of the same class.

  * Use of SGLT2 inhibitors or GLP-1 receptor agonists within 3 months prior to screening.
  * Adjustments to antidiabetic treatment regimens within 3 months prior to screening.
  * Hospitalization due to acute coronary syndrome (ST-segment elevation myocardial infarction, non-ST-segment elevation myocardial infarction, or unstable angina), percutaneous coronary intervention, or cardiac surgery within 30 days prior to the screening visit.
  * Volume depletion.
  * Chronic (>2 weeks) systemic glucocorticoid therapy or use of glucocorticoids within 4 weeks prior to screening (except for topical, intraocular, intranasal, or inhaled administration).
  * Pregnancy, lactation, or plans for pregnancy within the next 6 months.
  * Persistently elevated serum transaminase levels (more than 3 times the upper limit of normal).
  * Renal impairment (estimated glomerular filtration rate [eGFR] < 45 mL/min/1.73 m²).
  * History of malignant tumors.
  * Presence of acute complications (e.g., ketoacidosis, diabetic ketoacidosis, lactic acidosis, or hyperosmolar coma).
  * Systemic autoimmune diseases, such as systemic lupus erythematosus.
  * Clinically significant urinary tract infections and/or genital infections, or a history of recurrent urinary tract and/or genital infections.
  * Any other factors deemed by the investigator to potentially affect the efficacy or safety evaluation of the study.
  * Participation in other clinical trials and receipt of investigational drugs within 3 months prior to screening.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the mean amplitude of glycemic excursions at 16 weeks | From enrollment to the end of treatment at 16 weeks

SECONDARY OUTCOMES:
Change from Baseline in the immunophenotype of peripheral blood mononuclear cells at 16 weeks | From enrollment to the end of treatment at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Qing Su, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiaotong University School of Medicine, Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No